CLINICAL TRIAL: NCT03977428
Title: Central China Congenital Heart Disease Associated Pulmonary Arterial Hypertension Cohort Study
Acronym: CHD-PAHCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019LMC-1
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: standard of care — No intervention, this a patient registry and is purely an observational study

SUMMARY:
The study will recruit and follow up patients for five years patients newly diagnosed with congenital heart disease associated pulmonary arterial hypertension(CHD-PAH) from the investigator's hospital. The main aim of the study is to describe the aetiology, natural history and management practices of CHD-PAH in central China.

DETAILED DESCRIPTION:
baseline include: An echocardiogram to assess the size, shape, pumping action and the extent of any damage to the heart.

Lung function tests which include blowing measurements to assess gas volumes within the lungs as well as assessment of how the lungs exchange gases.

Right heart catheterisation (RHC) to diagnose PAH Optional Cardiac Magnetic Resonance tests. 6 minute walk distance (6MWD). To measure exercise capacity Electrocardiogram (ECG), a test that measures the electrical activity of the heart Blood tests

main outcome measure include:

death heart/lung transplantation atrial septostomy hospitalization due to worsening of PAH start of new specific PAH treatment persistent decrease of >15% from baseline in 6MWD (or >30% compared with last study-related measurement) persistent worsening of World Health Organization (WHO) Functional Class (FC）

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of CHD-PAH (by RHC)

Exclusion Criteria:

* PAH due to other criteria;
* unable to participate

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with diagnosis of CHD-PAH
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
survival | 5 years
  To recruit a cohort of CHD-PAH cases. define the death as the primary outcome

SECONDARY OUTCOMES:
clinical worsening | 5 years
  number of patients were dead, or having heart/lung transplantation, atrial septostomy, hospitalization due to worsening of PAH, starting of new specific PAH treatment, persistent decrease of >15% from baseline in 6MWD (or >30% compared with last study-related measurement), persistent worsening of WHO FC

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Qiu, Principal Investigator — Wuhan Asian Heart Hospital
Locations (1):
- Wuhan Asian Heart Hospital, Wuhan, China

IPD SHARING:
Plan to Share IPD: No